CLINICAL TRIAL: NCT00128583
Title: Response of In-Transit Melanoma to Systemic Treatment With the Specific Active Immunotherapeutic Agent, Canvaxin™
Brief Title: Vaccine Therapy in Treating Patients With Malignant Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CancerVax Corporation (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000439529; CV-MMAIT-5-001
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2005-09

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — Canvaxin

INTERVENTIONS:
Biological: polyvalent melanoma vaccine

SUMMARY:
RATIONALE: Vaccines made from tumor cells may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase II trial is studying vaccine therapy to see how well it works in treating patients with malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response in patients with in-transit cutaneous malignant melanoma treated with active immunotherapy comprising polyvalent melanoma vaccine (Canvaxin™).

OUTLINE: This is an open-label, multicenter study.

Patients receive polyvalent melanoma vaccine (Canvaxin™) subcutaneously to the armpit and groin areas every 2 weeks for approximately 10 weeks (5 doses) and then every 4 weeks for up to approximately 1 year of total treatment (total of 15 doses). Patients with no evidence of response at week 24 receive no further treatment. Patients whose disease continues to respond after completion of study treatment are eligible for a new study in which they will continue treatment with polyvalent melanoma vaccine (Canvaxin™).

After completion of study treatment, patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma
* At least 1 in-transit skin lesion measuring 3-10 mm in the longest diameter

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-07

PRIMARY OUTCOMES:
Response

CONTACTS AND LOCATIONS:
Overall Officials: Linda Strause, Study Chair — CancerVax Corporation
Locations (11):
- United States (9):
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - John Wayne Cancer Institute at Saint John's Health Center, Santa Monica, California
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - CCOP - Dayton, Dayton, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Simmons Cancer Center at University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
- Australia (2):
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland